CLINICAL TRIAL: NCT04295967
Title: Vasculogenic Mimicry in Urothelial Carcinoma and Its Association With Clinicopathologic Features
Brief Title: Vasculogenic Mimicry in Urothelial Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ereny Kamal Louis, administrator, Assiut University
Other Study IDs: VM in urothelial carcinoma
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: presence of recurrence of urothelial carcinoma
  Interventions: Other: formalin fixed paraffin embedded blocks
- 2: absence of recurrence of urothelial carcinoma
  Interventions: Other: formalin fixed paraffin embedded blocks

INTERVENTIONS:
Other: formalin fixed paraffin embedded blocks — The study will be conducted using formalin fixed paraffin embedded blocks of seventy cases of urothelial carcinomas .CD31-PAS dual-staining will be performed to confirm the presence of VM.

SUMMARY:
In this study, the investigators aim at:

1. Evaluate the presence of vasculogenic mimicry in urothelial carcinomas by CD31-PAS double staining.
2. Correlate the presence of vasculogenic mimicry with the clinicopathologic features as age, sex, TNM stage, pathological grade, recurrence, carcinoma in situ, lymphovascular emboli, lymph node metastasis, necrosis, surgical margin, multifocality and tumor size in urothelial carcinoma.

DETAILED DESCRIPTION:
Bladder cancer is the ninth most common cancer worldwide which seriously affects human health. In Egypt, it is the third common malignant tumor.

Urothelial carcinoma (UC) is considered the most common histologic type of bladder cancer.

It is well recognized that the biological behavior of several cancers is closely related to their blood supply. Tumor progression and metastasis have been long associated with tumor angiogenesis. However, several studies demonstrated that vascular targeting drugs which induce endothelial cell apoptosis have a little effect. So, it has been suggested that novel tumor microcirculation patterns may exist in these neoplasms.

Vasculogenic mimicry (VM), is a novel tumor microcirculation system. Maniotis et al initially discovered VM in melanoma and defined these channels to be composed of tumor basement membrane lined externally by tumor cells, lacking blood vessel endothelium and containing plasma and red blood cells. So VM can be distinguished using immunohistochemical (IHC) staining and histochemical double staining. VM is CD31- or CD34-negative (endothelial markers) and periodic acid-Schiff (PAS) positive.

Vasculogenic mimicry was detected in several malignant tumors. Several studies reported that VM can promote tumor progression and metastasis and it is positively associated with pathological grade, stage, recurrence and drug resistance. Previous studies which evaluate, the role of VM in urothelial carcinoma yield controversial results. So, the value of VM in urothelial carcinomas and its relation to the clinicopathologic parameters remains to be elucidated.

ELIGIBILITY:
Inclusion Criteria:

* - Specimens of urothelial carcinoma.

Exclusion Criteria:

* - Any criteria that not fulfill the inclusion criteria such as resected urinary bladder tumors other than urothelial carcinoma.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted using formalin fixed paraffin embedded blocks of sixty cases of urothelial carcinomas . These blocks will be obtained from laboratory archives of the Pathology Department, Assiut University Hospital, Faculty of Medicine. Clinical data for this study will be obtained from laboratory archives of the pathology department, Assiut University Hospital, Assiut University.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Evaluate the presence of vasculogenic mimicry in urothelial carcinomas by CD31-PAS double staining | baseline

SECONDARY OUTCOMES:
Correlate the presence of vasculogenic mimicry with the clinicopathologic features in urothelial carcinoma. | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Abeer R Mohamed, professor, Principal Investigator — Assiut University

REFERENCES:
- [Background] Zhou L, Chang Y, Xu L, Hoang ST, Liu Z, Fu Q, Lin Z, Xu J. Prognostic value of vascular mimicry in patients with urothelial carcinoma of the bladder after radical cystectomy. Oncotarget. 2016 Nov 15;7(46):76214-76223. doi: 10.18632/oncotarget.12775. PMID 27776348
- [Background] Aso Y, Ushiyama T, Suzuki K, Tajima A, Naide Y, Ohshima S, Matsuura O, Fukushima M, Ota K, Ono Y, et al. [Use of VM-26 as a single agent in the treatment of transitional cell carcinoma of the urinary tract]. Nihon Gan Chiryo Gakkai Shi. 1988 May 20;23(5):1046-51. No abstract available. Japanese. PMID 3418215